CLINICAL TRIAL: NCT04911296
Title: Pill Swallow Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RANI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP-0003
Record Dates: First submitted 2021-05-27; First posted 2021-06-03 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Not Determined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Swallow Group (Other)
  Interventions: Other: Mock-RP

INTERVENTIONS:
Other: Mock-RP — Standard 000 capsule filled with potato starch, enteric-coated with colorant and lubricious coating.

SUMMARY:
A prospective, single-center, open-label, single-arm, observational study assessing participant experience with swallowing the Mock-RP

ELIGIBILITY:
Inclusion Criteria:

1. Participant age is 21 - 75 years
2. Participant understands the nature of the study, is willing to comply with protocol defined evaluations, and provide written informed consent
3. Participant currently taking injections to treat a chronic disorder
4. Non-pregnant, non-lactating female NOTE: Females who are of childbearing potential must have had a negative pregnancy test on day of screening

Exclusion Criteria:

1. Active case of COVID-19
2. History of Dysphagia
3. History of dementia (e.g., Alzheimer's, vascular dementia, dementia with Lewy bodies, etc.)
4. Participant self-reports issues with swallowing pills.
5. History of drug or alcohol abuse or any other factor that, in the Investigator's opinion, may interfere with the participant's ability to cooperate and comply with the study procedures
6. History of allergic reaction to a component of the Mock-RP
7. History which, in the investigator's judgement, makes the participant ineligible or exposes the participant to unacceptable risks

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials of Texas, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Swallow Group
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Swallow Group
Number analyzed (Participants) | 150
Age, Customized [Count of Participants; unit: Participants]
  21 - 50 years | 50
  51 - 65 years | 50
  66 - 75 years | 50
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex stratified by age groups.
  Participants
    21 - 50 years: number analyzed (Participants) | 50
    21 - 50 years: Female | 29
    21 - 50 years: Male | 21
    51 - 65 years: number analyzed (Participants) | 50
    51 - 65 years: Female | 28
    51 - 65 years: Male | 22
    66 - 75 years: number analyzed (Participants) | 50
    66 - 75 years: Female | 28
    66 - 75 years: Male | 22
    Total: Female | 85
    Total: Male | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race stratified by age groups
  Participants
    21 - 50 years: number analyzed (Participants) | 50
    21 - 50 years: Black - Non-Hispanic | 6
    21 - 50 years: American Indian/Alaskan Native | 1
    21 - 50 years: Hispanic | 32
    21 - 50 years: Asian/Pacific Islander | 0
    21 - 50 years: White - Non-Hispanic | 11
    51 - 65 years: number analyzed (Participants) | 50
    51 - 65 years: Black - Non-Hispanic | 5
    51 - 65 years: American Indian/Alaskan Native | 1
    51 - 65 years: Hispanic | 28
    51 - 65 years: Asian/Pacific Islander | 0
    51 - 65 years: White - Non-Hispanic | 16
    66 - 75 years: number analyzed (Participants) | 50
    66 - 75 years: Black - Non-Hispanic | 7
    66 - 75 years: American Indian/Alaskan Native | 0
    66 - 75 years: Hispanic | 24
    66 - 75 years: Asian/Pacific Islander | 2
    66 - 75 years: White - Non-Hispanic | 17
    Total: Black - Non-Hispanic | 18
    Total: American Indian/Alaskan Native | 2
    Total: Hispanic | 84
    Total: Asian/Pacific Islander | 2
    Total: White - Non-Hispanic | 44
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 150
BMI [Mean (Full Range); unit: kg/m^2] — Population: BMI stratified by age groups
  kg/m^2
    21 - 50 years: number analyzed (Participants) | 50
    21 - 50 years | 35.54 [20.6 to 61.6]
    51 - 65 years: number analyzed (Participants) | 50
    51 - 65 years | 34.87 [18.5 to 51.9]
    66 - 75 years: number analyzed (Participants) | 50
    66 - 75 years | 32.93 [18.7 to 47.8]
    Total | 34.45 [18.5 to 61.6]

OUTCOME MEASURES:

1. Primary Outcome: Successful Swallowing of the Mock-RP
Description: Percent of participants successfully swallowing the Mock-RP as reported on the questionnaire.
Time Frame: Immediately after swallowing
Measure: Count of Participants; unit: Participants
Arm/Group | Swallow Group
Number analyzed (Participants) | 150
Participants | 150

2. Primary Outcome: Percent of Participants Who Would Chose a Pill Instead of Injection
Description: Assess if a participant would choose a pill instead of their current injection therapy if a pill becomes available.
Time Frame: Immediately after swallowing
Measure: Count of Participants; unit: Participants
Arm/Group | Swallow Group
Number analyzed (Participants) | 150
Participants | 136

3. Primary Outcome: Mock-RP Swallowing Experience
Description: Participant experience with swallowing Mock-RP stratified by number of years using injections.
Time Frame: Immediately after swallowing
Measure: Count of Participants; unit: Participants
Groups:
- <1 Year; 1-5 Years; >5 Years: How long have you been taking injections for your condition?
Arm/Group | <1 Year | 1-5 Years | >5 Years
Number analyzed (Participants) | 16 | 59 | 75
Participants
  Easy | 12 | 46 | 56
  Large Pill - Easy | 3 | 8 | 14
  Challenging Due to Size | 1 | 3 | 4
  No Comment | 0 | 2 | 1
Statistical Analysis 1: Comparison: <1 Year vs 1-5 Years vs >5 Years; Test type: Other; p = 0.935, Fisher Exact

4. Primary Outcome: Mock-RP Swallowing Experience
Description: Participants' experience with swallowing Mock-RP was stratified by age (21-50, 51-65, 66-75 years).
Time Frame: Immediately after swallowing
Measure: Count of Participants; unit: Participants
Groups:
- 21 - 50 Years; 51 - 65 Years; 66 - 75 Years: Age at time of enrollment.
Arm/Group | 21 - 50 Years | 51 - 65 Years | 66 - 75 Years
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Easy | 36 | 37 | 41
  Large Pill - Easy | 10 | 9 | 6
  Challenging Due to Size | 4 | 3 | 1
  No Comment | 0 | 1 | 2
Statistical Analysis 1: Comparison: 21 - 50 Years vs 51 - 65 Years vs 66 - 75 Years; Test type: Other; p = 0.536, Fisher Exact

5. Primary Outcome: Mock-RP Swallowing Experience
Description: Participants completed a questionnaire after swallowing the Mock-RP stating if they would select a pill alternative over their current injections - stratified by frequency of injection treatment.
Time Frame: Immediately after swallowing
Measure: Count of Participants; unit: Participants
Groups:
- Daily; Every 2 Weeks; Weekly; Monthly: Injection Frequency
Arm/Group | Daily | Every 2 Weeks | Weekly | Monthly
Number analyzed (Participants) | 102 | 2 | 36 | 10
Participants
  No | 10 | 0 | 2 | 2
  Yes | 92 | 2 | 34 | 8

6. Primary Outcome: Adverse Events
Description: All adverse events categorized by type and frequency.
Time Frame: Immediately after swallowing
Measure: Count of Participants; unit: Participants
Arm/Group | Swallow Group
Number analyzed (Participants) | 150
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Swallow Group
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT04911296/Prot_SAP_000.pdf